CLINICAL TRIAL: NCT04174651
Title: The Cerebral Mechanism of Stress-Induced Spontaneous Scratching in Healthy Volunteers and Patients With Atopic Dermatitis (AD)
Brief Title: Stress-induced Scratching in Healthy and AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hideki Mochizuki, Assistant Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20190833
Record Dates: First submitted 2019-10-10; First posted 2019-11-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Healthy; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: Crossover randomization within the arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with AD with MRI (Experimental): Participants that are diagnosed with AD will receive both the acute stress condition (TSST) and the control condition (watching a landscape video). The order when the 2 conditions will be provided is randomized per participant and completed 2 weeks apart. These subjects will be evaluated with MRI.
  Interventions: Behavioral: Trier Social Stress Test (TSST); Behavioral: Landscape Video
- Healthy Participants with MRI (Experimental): Healthy participants will receive both the acute stress condition (TSST) and the control condition (watching a landscape video). The order when the 2 conditions will be provided is randomized per participant and completed 2 weeks apart. These subjects will be evaluated with MRI.
  Interventions: Behavioral: Trier Social Stress Test (TSST); Behavioral: Landscape Video

INTERVENTIONS:
Behavioral: Trier Social Stress Test (TSST) — Participants randomized to receive the acute stress condition will undergo the TSST wherein the participant will be introduced to an upcoming task (i.e., job interview) and allowed to prepare (2 minutes). The participant will then be required to speak (job interview) for 4 minutes in front of 2 experimenters. After completion of the interview, participants will be asked to perform a mental arithmetic task for 4 minutes.
Behavioral: Landscape Video — Participants randomized to receive the control condition will be watching a landscape video for 10 minutes.

SUMMARY:
The purpose of this study is to examine scratching behavior and identify brain areas responsible for stress-induced spontaneous scratching in patients with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects and AD patients between 18 and 59 years of age.
2. Healthy subjects: In general, good health without history of neurological and psychiatric diseases.
3. AD patients: An average itch rating of 3 out of 10 or greater in the past two weeks using a Numerical Rating Scale (NRS).
4. All patients will be required to cease use of oral antihistamines from the night before each study visit until the end of the experiment. The purpose is to avoid that participants fall asleep during MRI measurement due to side effect oral antihistamine (i.e., sedation).
5. Women of child bearing potential will be administered a pregnancy test to verify that they are not pregnant.
6. MRI Compatibility, criteria include having no major contraindication for MRI (pacemaker, vascular stents, metallic ear tubes, and absence of metal implants or braces) as assessed by MRI technologist using site approved screening form.
7. Participants have to be able to speak and read English fluently.
8. Participants must have signed a written informed consent before being enrolled in the study

Exclusion Criteria:

1. Individuals under 18 or over 59 years of age.
2. Inability to complete the required measures.
3. Suffering from any disease state or physical condition, which would increase their health risk by study participation.
4. Currently enrolled in any investigational study in which the subject is receiving any type of drug, biological, or non-drug therapy.
5. Recent initiation (within last 3 months) of centrally acting agents such as antidepressants, neuroleptics or neuropathic medications.
6. Patients who use centrally acting agents only when they need. The purpose is to avoid a risk of acute effect of these agents on brain activity and perceived stress due to the stress task.
7. Current treatment with opioid analgesics.
8. Uncontrolled thyroid disease.
9. Use of illicit drugs or history of opiate addiction.
10. Diagnosis of a major psychiatric disorder such as schizophrenia, major depression or bipolar disorder that is active right now.
11. Any known diseases or disorders that may affect conducting the experiments (e.g., intracranial pathology, claustrophobia, severe respiratory or cardiovascular problems, active fibromyalgia) or diseases that have potential risks of infections (e.g., HIV, Hepatitis C, etc).
12. Inability to speak and read English.
13. Being pregnant.
14. Incarcerated.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Changes in brain activity | Baseline, 15 minutes
  Changes in brain activity will be measured as change in Arterial spin Labeling (ASL) which reflects regional cerebral blood flow. This will be evaluated using functioning magnetic resonance imaging (fMRI).
Change in time of spontaneous scratching | Baseline, 15 minutes
  Change in spontaneous scratching for behavioral only arms will be calculated by subtracting total duration of scratching behavior before and after the TSST and Landscape video.

SECONDARY OUTCOMES:
Correlation of perceived stress with stress-induced brain activity | 60 minutes
  The correlation of stress-induced brain activity evaluated as ASL signals will be evaluated against participant's stress questionnaire scores and biological stress marker (saliva cortisol levels).

CONTACTS AND LOCATIONS:
Overall Officials: Hideki Mochizuki, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No